CLINICAL TRIAL: NCT05824390
Title: A Randomized, Controlled Clinical Study of Rituximab in Treatment of Primary IgA Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XIEJINGYUAN (Other)
Collaborators: Dongfang Hospital Affiliated to Tongji University (Other); Shanghai Pudong New Area People's Hospital (Other); Ruijin Hospital North Shanghai Jiao Tong University School of Medicine (Unknown); Ningbo Municipal Yinzhou District No.2 Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Xiamen Humanity Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor-Investigator, XIEJINGYUAN, professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RuijinHRIGA
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( ACEi and / or ARB + rituximab group ) (Experimental): Patients in the experimental group were treated with the maximum tolerable dose of angiotensin converting enzyme inhibitor ( ACEI ) and / or angiotensin II receptor blocker ( ARB ) combined with rituximab. The specific usage and dosage are as follows : On the basis of the use of ACEI and / or ARB, rituximab was used on D1 and D31 days, 1 g each time, intravenous drip, twice in total. Add 1 g rituximab at 6 months. All patients who received rituximab were given oral acetaminophen ( 1g ), diphenhydramine hydrochloride ( 50mg ) and intravenous methylprednisolone ( 40mg ) 30-60min before the beginning of infusion. ACEI and / or ARB were given daily maximum tolerable dose according to individual factors of subjects.
  Interventions: Drug: rituximab group
- Group B ( ACEi and / or ARB ) (No Intervention): According to the individual factors of the subjects, the maximum tolerable dose of angiotensin converting enzyme inhibitor ( ACEI ) and / or angiotensin II receptor blocker ( ARB ) were used daily.

INTERVENTIONS:
Drug: rituximab group — Rituximab is a human-mouse chimeric monoclonal antibody specifically targeting B cell surface antigen CD20. CD20 may act as a calcium channel to play a certain signal role and participate in the regulation of B cell maturation and differentiation. Once combined with CD20, RTX consumed CD20 + B fines through antibody-dependent cell-mediated cytotoxicity, complement-dependent cytotoxicity and direct induction of apoptosis. Recent studies have shown that B cell depletion therapy has a certain effect on many autoantibodies-mediated kidney diseases ( such as membranous nephropathy, lupus nephritis, etc. ). Therefore, rituximab combined with CD20 antigen on the surface of B cells can exhaust B cells that produce antibodies and play a therapeutic role by reducing antibody production, so this therapy also has potential therapeutic value for IgAN patients.
  Other Names: ACEi and / or ARB
  Arms: Group A ( ACEi and / or ARB + rituximab group )

SUMMARY:
A study to evaluate safety and activity in treatment of IgAN patients using Rituximab in combination with RASi(ACEI and/or ARB) compared with RASi.

DETAILED DESCRIPTION:
IgA nephropathy (IgAN, IgA nephropathy), is currently the most common glomerular disease worldwide, which is characterized by High population quantity, wide distribution, strong heterogeneity.

Diagnosis of Urinary protein control level within 1 year is one of the important predictors of renal failure in IgAN patients.Previous studies have shown that patients with renal insufficiency, hypertension, or urinary protein > 1g at 24h during renal biopsy, and those with poor urinary protein control within 1 year of follow-up, have a higher risk of disease progression, and more than 30-50% of patients will develop into end-stage renal disease (ESRD) within 10 years.

The recommended treatments for IgAN in the KDIGO guidelines include: RASi, glucocorticoid, immunosuppressor, antiplatelet drugs, lipid-lowering drugs, etc. Several trials have demonstrated the benefit of RASi in retarding disease progression in IgAN patients with proteinuria, but there is currently no specific treatment for IgAN.

In recent years, it has been found that excessive production of Galactos-deficient IgA1 is one of the initiating factors of the pathogenesis of IgAN. Infection by pathogenic microorganisms induces lymphocytes in IgAN patients to produce anti-GD-IgA1 autoantibodies (second strike), which forms circulating immune complexes to deposit in the kidney and activates complement, which is an important pathogenesis of IgAN.However, recent studies have suggested that B-cell depletion therapy is effective for many aabs mediated renal diseases (e.g., membranous nephropathy, lupus nephritis, etc.). Rituximab, which combined with CD20 antigen on the B cell surface, can deplete B cells and play a therapeutic role by reducing antibody production. Therefore, the treatment of rituximab has potential therapeutic value for IgAN patients as well.

However, there were very few studies which have shown the efficacy and safety of rituximab in the treatment of IgA nephropathy, only groups reported abroad, and the results were inconsistent. At present, there have been no randomized controlled studies to verify the safety and efficacy of rituximab in the treatment of IgA nephropathy, especially in Chinese with high incidence of IgAN.

In this study, treatment of rituximab combining with RASi will be compared with RASi for IgAN patients, to explore an effective and safer regimen for IgAN, so as to bring more hope to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, no gender limit;
2. Renal biopsy confirmed primary IgA nephropathy;
3. Assess glomerular filtration rate ( eGFR )>30ml/min/1.73m2 (calculated according to the CKD-EPI formula);
4. After 3 months of treatment with the maximum tolerated dose of ACEI and/or ARB, the following two points should be met:

1) 24hurinary protein ≥ 1g; 2) Blood pressure <130/80 mmHg; 5. Serum albumin> 25g/L; 6. Voluntarily sign the informed consent.

Note : It is suggested that active IgAN patients should be selected. Active IgAN is specifically defined as conforming to any of the following :

1. ) intradermal augmentation ( E1 ),
2. ) crescentic body 0 - 50 % ( C1 / C2 ),
3. ) fibrinoid necrosis,
4. ) more interstitial inflammatory cell infiltration. At the same time, the proportion of sclerosis was low ( spherical or segmental sclerosis ball < 50 % ), and interstitial fibrosis was low ( below T2 ).

Exclusion Criteria:

1. Glucocorticoid used for immunosuppressive therapy indications, such as : nephrotic syndrome, pathology for small lesions with IgA nephropathy. or the proportion of crescents confirmed by renal biopsy within 12 months was more than 50 %.
2. Clinically confirmed cirrhosis, chronic active liver disease or hepatitis B, hepatitis C or HIV can detect viral replication.
3. Clinically confirmed IgA nephropathy secondary to systemic diseases such as systemic lupus erythematosus, allergic purpura.
4. Patients with non-simple IgA nephropathy, such as diabetic nephropathy or obesity-related nephropathy.
5. A history of active systemic infection or severe infection occurred one month before enrollment.
6. Those who are pregnant or lactating or unwilling to take contraceptive measures.
7. Current or recent ( within 30 days ) exposure to any research drug. 8. Patients with allergic reactions to rituximab and / or known allergic reactions.
8. Patients with allergic reactions to rituximab and / or known allergic reactions.
9. Laboratory tests should be excluded if they meet the following standards :

(1) Hemoglobin <80g/L; (2) Platelets<80×109/L; (3) Neutrophils <1.0×109/L; (4) In addition to being related to the primary disease, aspartate aminotransferase (AST) or alanine aminotransferase (ALT)>2.5×upper limit of normal; 10. Continuous use of hormones or other immunosuppressive therapy in the past 6 months; 11. Accompanying or past malignant tumors, except for fully treated skin basal or squamous cell carcinoma or cervical carcinoma in situ; 12. History of psychosis may interfere with normal participation in this study; 13. Patients with major heart or lung diseases (including obstructive pulmonary disease); 14. In acute and chronic tuberculosis infection period (tuberculin test positive, chest X-ray suspected tuberculosis patients); 15. Patients with history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 16. Low weight (weight < 50kg) should be excluded; 17. Other investigators judged patients unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in proteinuria levels over 1 year compared with baseline | 1 year
  changes in proteinuria levels over 1 year compared with baseline

SECONDARY OUTCOMES:
The proportion of 50% reduction in mean urinary protein compared with baseline over 1 year | 1 year
  Statistical data of proportion of 50% reduction in mean urinary protein compared with baseline over 1 year
The proportion of 50% reduction in mean urinary protein compared with baseline over 6 months | 6 months
  Statistical data of proportion of 50% reduction in mean urinary protein compared with baseline over 6 months
Changes in proteinuria levels over 6 months compared with baseline | 6 months
  Changes in proteinuria levels over 6 months compared with baseline
Changes in eGFR levels over 1 year compared with baseline | 1 year
  changes in eGFR levels over 1 year compared with baseline
Changes of Gd-IgA1 levels | 1 year
  Changes of Gd-IgA1 levels
Incidence of adverse events | 1 year
  Incidence of adverse events
Incidence of ESRD | 1 year
  Incidence of ESRD
Proportion of eGFR decreased by 50 % or serum creatine doubled compared with baseline | 1 year
  Proportion of eGFR decreased by 50 % or serum creatinine doubled compared with baseline
Incidence rate of infection | 1 year
  Incidence rate of infection

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China